CLINICAL TRIAL: NCT05388825
Title: A Randomized, Double-blind, Placebo-controlled, Two-cohort, Three-way Crossover Clinical Trial to Evaluate the Pharmacodynamic Effect of Different Doses of TPN171H Tablets in Mild to Moderate Male Erectile Dysfunction
Brief Title: Pharmacodynamic Study of TPN171H Tablets in Patients With Mild to Moderate Erectile Dysfunction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vigonvita Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: TPN171H-E202
Record Dates: First submitted 2022-05-18; First posted 2022-05-24 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Sequence 1 (Experimental): N=14 subjects receive 2.5 mg TPN171H and 10 mg Placebo for Period 1; 5 mg TPN171H and 10 mg Placebo for Period 2 ; 10 mg Placebo and 5 mg Placebo for Period 3.
  Interventions: Drug: TPN171H 2.5mg; Drug: TPN171H 5mg; Drug: Placebo 5mg; Drug: Placebo 10mg
- Sequence 2 (Experimental): N=14 subjects receive 5 mg TPN171H and 10 mg Placebo for Period 1; 10 mg Placebo and 5 mg Placebo for Period 2 ; 2.5 mg TPN171H and 10 mg Placebo for Period 3.
  Interventions: Drug: TPN171H 2.5mg; Drug: TPN171H 5mg; Drug: Placebo 5mg; Drug: Placebo 10mg
- Sequence 3 (Experimental): N=14 subjects receive 10 mg Placebo and 5 mg Placebo for Period 1; 2.5 mg TPN171H and 10 mg Placebo for Period 2; 5 mg TPN171H and 10 mg Placebo for Period 3.
  Interventions: Drug: TPN171H 2.5mg; Drug: TPN171H 5mg; Drug: Placebo 5mg; Drug: Placebo 10mg
- Sequence 4 (Experimental): N=14 subjects receive 5 mg TPN171H and 10 mg Placebo for Period 1; 10 mg TPN171H and 5 mg Placebo for Period 2; 10 mg Placebo and 5 mg Placebo for Period 3.
  Interventions: Drug: TPN171H 5mg; Drug: TPN171H 10mg; Drug: Placebo 5mg; Drug: Placebo 10mg
- Sequence 5 (Experimental): N=14 subjects receive 10 mg TPN171H and 5 mg Placebo for Period 1; 10 mg Placebo and 5 mg Placebo for Period 2; 5 mg TPN171H and 10 mg Placebo for Period 3.
  Interventions: Drug: TPN171H 5mg; Drug: TPN171H 10mg; Drug: Placebo 5mg; Drug: Placebo 10mg
- Sequence 6 (Experimental): N=14 subjects receive 10 mg Placebo and 5 mg Placebo for Period 1; 5 mg TPN171H and 10 mg Placebo for Period 2; 10 mg TPN171H and 5 mg Placebo for Period 3.
  Interventions: Drug: TPN171H 5mg; Drug: TPN171H 10mg; Drug: Placebo 5mg; Drug: Placebo 10mg

INTERVENTIONS:
Drug: TPN171H 2.5mg — TPN171H 2.5mg is recommended to take warm water on an empty stomach (2 hours or more after dinner)
  Arms: Sequence 1; Sequence 2; Sequence 3
Drug: TPN171H 5mg — TPN171H 5mg is recommended to take warm water on an empty stomach (2 hours or more after dinner)
Drug: TPN171H 10mg — TPN171H 10mg is recommended to take warm water on an empty stomach (2 hours or more after dinner)
  Arms: Sequence 4; Sequence 5; Sequence 6
Drug: Placebo 5mg — Placebo 5mg is recommended to take warm water on an empty stomach (2 hours or more after dinner)
Drug: Placebo 10mg — Placebo 10mg is recommended to take warm water on an empty stomach (2 hours or more after dinner)

SUMMARY:
This study is a randomized, double-blind, placebo-controlled, two-cohort, three-cycle crossover (at least a 5-day cleaning period per cycle), and a multicenter clinical trial design.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled, two-cohort, three-cycle crossover (at least a 5-day cleaning period per cycle), and a multicenter clinical trial design. The pharmacodynamic effects of different doses of TPN171H tablets on mild to moderate male patients with erectile dysfunction were evaluated by penile plethysmography (RigiScan PlusTM technique) using audiovisual sexual stimulation (AVSS).

ELIGIBILITY:
Inclusion Criteria:

* 18 years to 65 years (inclusive)
* Males with ED at least 6 months, meets the diagnosis of mild and moderate erectile dysfunction，8≤IIEF-5 ≤ 21
* Patients who are willing to stay away from any other medicines or treatments for ED during this study period
* Patients (including partners) who are willing to take proper contraceptive during the study and within 3 months after the study completed
* Patients who have voluntarily decided to participate in this study, and signed the informed consent form

Exclusion Criteria:

* Patients who have a history of hypersensitivity to other PDE5 inhibitors or TPN171H
* Patients with anatomical malformations of the penis
* Patients with primary hypoactive sexual desire
* Patients with ED, which is caused by any other primary sexual disorder
* Patients with ED ,which is caused by spinal injury or have had a radical prostatectomy or other surgery
* Patients who have a penile implant
* Patients who have not responded to PDE5 inhibitors or who have an adverse reaction leading to discontinuation
* CYP3A4 potent inhibitors, potent inducers, and moderate inducers (except topical drugs) should be used within 28 days before the start of treatment or during the trial period
* Subjects who are taking nitrate or NO donor drugs, anti-androgens, guanylate cyclase agonists, or other drugs or treatments for the treatment of ED and cannot be discontinued
* Patients with the following cardiovascular disease:

Myocardial infarction or shock, or life-threatening arrhythmia within the last 6 months; Unstable angina or angina occurring during sexual intercourse within the last 3 months; Received coronary artery bypass grafting or percutaneous coronary intervention within the last 3 months；New York Heart Association Class 2 or greater heart failure in the last 6 months

* Uncontrolled hypotension (<90/60mmHg), uncontrolled hypertension(≥160/95mmHg)
* Diabetic patients whose FBS is over 1.5 fold of normal value, or whose HbA1c >9%, or with diabetes complications, such as diabetic nephropathy, peripheral neuropathy
* Patients with hepatic or renal dysfunction as per the following: AST, ALT>2*ULN, serum creatinine exceeds 20% of the upper limit of normal value
* Patients with active gastrointestinal ulcers and bleeding disorders
* Patients who have a history of NAION, or with a known genetically degenerative retinopathy, including retinitis pigmentosa
* Patients who have a history of sudden decrease or loss of hearing
* Patients with a history of severe central nervous system injury or peripheral muscular neurological disease in the past 6 months
* Patient with a history of malignancy
* Patients with significant neurological abnormalities
* Patients with alcohol addiction
* Patients with persistent abuse of drugs of dependence
* Patients who have a childbirth plan during the trial period and within 3 months after the trial
* Patients who are participating in the past 3 months from any other clinical trial (except those who have participated in the clinical trials of this product before)
* For other reasons besides the aforementioned cases, patient whose participation is deemed inappropriate due to clinically significant findings according to the medical decision of the principal investigator or the study personnel.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-01-04 (Actual); Study Completion 2023-02-17 (Actual)

PRIMARY OUTCOMES:
Duration of penile erections of greater than or equal to 60% rigidity as assessed by penile plethysmography (RigiScan PlusTM). | Baseline and during audiovisual sexual stimulation（60minutes）

SECONDARY OUTCOMES:
The starting time of penile erections of greater than or equal to 60% rigidity | Baseline and during audiovisual sexual stimulation（60minutes）
Duration of penile erections of greater than or equal to 60% rigidity as assessed by penile plethysmography (RigiScan PlusTM). | Baseline and during audiovisual sexual stimulation（minutes）
Percentage increase in penile enlargement | Baseline and during audiovisual sexual stimulation（60minutes）
The incidence of penile erection rigidity grade ≥ grade III. | Baseline and during audiovisual sexual stimulation（60minutes）

CONTACTS AND LOCATIONS:
Overall Officials: Hui Jiang, Principal Investigator — Peking University Third Hospital
Locations (8):
- China (8):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Henan Provincial People's Hospital, Zhenzhou, Henan
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jinlin
  - The Second Hospital of Dalian Medical University, Dalian, Liaoning

IPD SHARING:
Plan to Share IPD: No